CLINICAL TRIAL: NCT02783456
Title: The Influence of Aircraft Noise Exposure on Renal Hemodynamic in Healthy Individuals
Acronym: LÄRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CRCLÄRM2016
Record Dates: First submitted 2016-04-27; First posted 2016-05-26 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Healthy Individuals; Arterial Hypertension
Keywords: renal hemodynamic; central hemodynamic; pilot study; flight noise; healthy participant; renal plasma flow; filtration fraction; renal vascular resistance; calculated intra glomerular pressure
MeSH Terms: conditions — Hypertension | interventions — Noise; SIR1 protein, S cerevisiae

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Noise and silence (Active Comparator): Exposition of 80dB flight noise for 30 minutes and 30 minutes silence.
  Interventions: Procedure: Noise; Procedure: Silence
- silence and noise (Active Comparator): Exposition of 30 minutes silence.and 80dB flight noise for 30 minutes
  Interventions: Procedure: Noise; Procedure: Silence

INTERVENTIONS:
Procedure: Noise — The patient is exposed 30 min to the first sound pattern and during the renal hemodynamics will be measured. The following is a 1-hour break.
Procedure: Silence — The patient is exposed 30 min to the second sound pattern and during the renal hemodynamics will be measured.

SUMMARY:
Epidemiological studies have found a link between aircraft noise exposure and increased incidence of arterial hypertension and thus cardiovascular disease. The underlying pathophysiological mechanisms are not yet fully understood. The kidney acts as a long-term regulator of blood pressure and controls the extracellular sodium and water balance. Significant renal mechanisms of blood pressure regulation are the renin angiotensin system, renal sympathetic activity and sodium excretion. Animal work and clinical studies show that mental stress affects the renal plasma flow and urinary sodium excretion. The investigators observed a lower sodium excretion in situations of mental stress in subjects at risk for developing arterial hypertension. In healthy volunteers, a 30-minute mental stress test resulted in increased glomerular filtration rate, filtration fraction and an increase in urinary sodium excretion. In this pilot study the investigators analyzed the influence of 30 minutes standardized aircraft noise on renal and central hemodynamics.

DETAILED DESCRIPTION:
The World Health Organisation (WHO) estimates that (about 340 million population) 1 million annually health life years are lost by environmental noise exposure in high-income countries of Western Europe. Aircraft noise is thereby assessed at comparable volume as unpleasant as road and rail noise. Epidemiological studies have found a link between aircraft noise exposure and increased incidence of arterial hypertension and thus cardiovascular disease. The underlying pathophysiological mechanisms are not yet fully understood.

The kidney acts as a long-term regulator of blood pressure and controls the extracellular sodium and water balance. Significant renal mechanisms of blood pressure regulation are the renin angiotensin system, renal sympathetic activity and sodium excretion. Animal work and clinical studies show that mental stress affects the renal plasma flow and urinary sodium excretion. In spontaneously hypertensive rats environmental stress resulted in sodium retention, triggered by increased renal sympathetic nerve activity, which is the development of arterial hypertension. In a pilot study in subjects at risk for developing arterial hypertension, the investigator observed a lower sodium excretion by mental stress. In healthy volunteers, a 30-minute mental stress test resulted in increased glomerular filtration rate, filtration fraction and an increase in urinary sodium excretion.

In the rabbit noise exposure leads to an increase of frequency and amplitude of discharges of renal sympathetic nerve activity and accompanied by a reduction of renal plasma flow. The impact of aircraft noise on renal plasma flow and urinary sodium excretion has, to our knowledge, so far not been studied in humans.

In this pilot study the Clinical Research Center investigate the influence of 30 minutes standardized aircraft noise on renal hemodynamics.

Hemodynamic renal changes should be considered in the context of the systemic circulation. Therefore, the central hemodynamics is determined in the present pilot study by bioimpedance cardiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild-moderate arterial hypertension (grade 1-2)
* Informed consent in writing available
* Willing and able to comply with all requirements of the study
* Male, between 18 and 50 years (inclusive)
* Body Mass Index (BMI) 18-27 kg/m2
* Non-smoker
* Good general health as judged by the Investigator, as determined by medical history, physical examination, vital signs (systolic and diastolic blood pressure and pulse rate) and clinical laboratory parameters (clinical chemistry, hematology, and urinalysis).

Minor deviations of laboratory values, ECG, and vital sign parameters from the normal range may be accepted, if judged by the Investigator to have no clinical relevance.

Additional inclusion criteria for the cohort with arterial hypertension:

- uncomplicated arterial hypertension WHO grade 1-2, office blood pressure 140-179/90-109 mmHg

Exclusion Criteria for healthy individuals:

* Clinically significant abnormalities in physical examination, vital signs or clinical laboratory parameters (according to the Investigator's judgement).
* S-GOT or S-GPT levels > 2-times above the upper limit of normal range.
* eGFR < 60 ml/min/1,73m2 or kidney stones
* Clinically significant history of cardiovascular disease or any known present cardiovascular disease.
* History of clinically significant neurological, gastrointestinal, renal, hepatic, psychological, pulmonary, metabolic, endocrine, hematological, or other major disorders.
* Office blood pressure at screening higher than 140/100 mmHg
* Office heart rate at screening outside the range of 50-99 beats per minute (inclusive).
* Regular intake of medication within 1 month prior to study inclusion
* Participation in any other clinical study within 30 days prior to inclusion in this study.
* Clinically significant diseases (as judged by the investigator) within four weeks prior to screening
* History of alcohol or drug abuse.

Exclusion criteria for patients with arterial hypertension:

* Regular intake of medication within 1 month prior to study inclusion
* office blood pressure at screening visit > 180/110 mmHg
* secondary hypertension application of
* antihypertensive medication within 14 days prior to study inclusion
* of "other" medication
* Clinically significant abnormalities in physical examination, vital signs or clinical laboratory parameters (according to the Investigator's judgement).
* S-GOT or S-GPT levels > 2-times above the upper limit of normal range.
* eGFR < 60 ml/min/1,73m2 or kidney stones
* Clinically significant history of cardiovascular disease or any known present cardiovascular disease other than arterial hypertension.
* History of clinically significant neurological, gastrointestinal, renal, hepatic, psychological, pulmonary, metabolic, endocrine, hematological, or other major disorders, other than arterial hypertension.
* Office heart rate at screening outside the range of 50-99 beats per minute (inclusive).
* Regular intake of medication within 1 month prior to study inclusion
* Participation in any other clinical study within 30 days prior to inclusion in this study.
* Clinically significant diseases (as judged by the investigator) within four weeks prior to screening, other than arterial hypertension.
* History of alcohol or drug abuse.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
change in renal plasma flow (l/min) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roland E. Schmieder, Prof. Dr., Principal Investigator — University of Erlangen-Nürnberg Medical School
Locations (1):
- University of Erlangen-Nuremberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] A. Jumar, C. Ott, J.M. Harazny, K. Striepe, M.V. Karg, R.E. Schmieder. NEW MODEL TO INVESTIGATE THE INFLUENCE OF AIRCRAFT NOISE IN THE PATHOPHYSIOLOGICAL CONCEPT OF HYPERTENSION J Hypertens 2017;35, e-Supplement 2:e214 PP.15.32
- [Derived] Bosch A, Rauh M, Striepe K, Schiffer M, Schmieder RE, Kannenkeril D. Renal adaptation in pre-obesity patients with hypertension. J Hypertens. 2024 Nov 1;42(11):1958-1965. doi: 10.1097/HJH.0000000000003821. Epub 2024 Jul 19. PMID 39248112